CLINICAL TRIAL: NCT03111121
Title: Use of Sugammadex for Reversal of Paralysis in Microlaryngoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1610312153
Record Dates: First submitted 2017-03-23; First posted 2017-04-12 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Microlaryngoscopy; Rigid Bronchoscopy
Keywords: deeply anesthetized; ideal surgical exposure; muscle relaxation; Adults
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: Group 1: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6-1.2 mg/kg (vitals maintained within 20% of baseline). Group 1 will receive reversal with neostigmine (0.04 mg/kg and glycopyrrolate (0.01 mg/kg)
  Group 2: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6 -1.2 mg/kg (vitals maintained within 20% of baseline). Group 2 will receive reversal with sugammadex 4mg/kg
Who Masked: Care Provider
Masking Description: SINGLE BLIND: The nurses in PACU will be the only evaluators of the subject who will be blinded to the two groups. The PACU nurses will evaluate ALDRETE discharge criteria and make a note in the electronic medical records for the subject discharge time from PACU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Reversal of Paralysis in Microlaryngoscopy procedures: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6-1.2 mg/kg (vitals maintained within 20% of baseline). Standard anti-nausea prophylaxis - Ondansetran and Decadran intraoperative.After induction; amount of inhaled anesthetic and remifentanil used will be titrated based on hemodynamic parameters (maintained within 20% from baseline) and a BIS monitor.TOF testing done every 5 minutes:Group 1 will receive reversal with neostigmine (0.04 mg/kg and glycopyrrolate (0.01 mg/kg)
  Interventions: Drug: neostigmine; Drug: glycopyrrolate
- Group 2 (Active Comparator): Reversal of Paralysis in Microlaryngoscopy procedures: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6-1.2 mg/kg (vitals maintained within 20% of baseline). Standard anti-nausea prophylaxis - Ondansetran and Decadran intraoperative.After induction; amount of inhaled anesthetic and remifentanil used will be titrated based on hemodynamic parameters (maintained within 20% from baseline) and a BIS monitor.TOF testing done every 5 minutes: Group2 will receive reversal with sugammadex 4mg/kg
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — receive reversal with sugammadex 4mg/kg
  Arms: Group 2
Drug: neostigmine — receive reversal with neostigmine 0.04 mg/kg
  Arms: Group 1
Drug: glycopyrrolate — receive reversal with glycopyrrolate (0.01 mg/kg)
  Arms: Group 1

SUMMARY:
Use of Muscle relaxant and reversal with Sugammadex at end of airway procedures will reduce the time to extubation after end of procedure

DETAILED DESCRIPTION:
This is a prospective, clinical interventional, randomized single blinded single center study.

Hypotheses:

Primary Hypothesis: Use of Muscle relaxant and reversal with Sugammadex at end of airway procedures will reduce the time to extubation after end of procedure

Secondary Hypotheses:

Surgeon will report optimal surgical conditions for ease of exposure

Have less hemodynamic changes in the OR and PACU. ∆ in BP, HR and CO2 from base-line and incidence /frequency of 20% change in BP from baseline vitals (baseline= pre-induction vitals)

Decrease the amount of inhaled anesthetics

Decreased narcotics needed intra-operatively and post operatively

Decrease the total OR time

Subjects will meet ALDRETE PACU discharge criteria quicker in the PACU

Subject will have less adverse events and severe adverse events such as - hypotension, arrhythmia, hypoxia, stridor and re-intubation.

We note that the nurses in PACU will be blinded to whether the subjects were in Group 1 or 2.

Group 1: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6-1.2 mg/kg (vitals maintained within 20% of baseline). Group 1 will receive reversal with neostigmine (0.04 mg/kg and glycopyrrolate (0.01 mg/kg)

Group 2: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6 -1.2 mg/kg (vitals maintained within 20% of baseline). Group 2 will receive reversal with sugammadex 4mg/kg

Both groups will receive standard anti-nausea prophylaxis - Ondansetran and Decadran intraoperative.

After induction, the amount of inhaled anesthetic and remifentanil used will be titrated based on hemodynamic parameters (maintained within 20% from baseline) and a BIS monitor.

All subjects will have TOF testing done every 5 minutes throughout the procedure and tabulated in the Electronic Medical Record (EMR).

At the end of the procedure patient will be extubated when the subject meets the following criteria:

Tidal volume : > 5 cc /Kg Respiratory rate: >8 /min O2sat > 95% ON 100% inspired oxygen

With vitals at 20% of baseline. Extubation will begin when the surgeon states, "We are done". This usually coincides with the withdrawal of the scope. The start and end times for extubation will be recorded in the Electronic Medical Record.

The PACU nurses will evaluate ALDRETE discharge criteria and make a note in the electronic medical records for the subject discharge time from PACU. The nurses in PACU will be the only evaluators of the subject who will be blinded to the two groups

ELIGIBILITY:
Inclusion Criteria:

Microlaryngoscopy or rigid bronchoscopy for vocal cord and tracheal procedures

Age 18 years or older,

ASA physical status I-III

Ability to give written informed consent.

Exclusion Criteria:

Known or suspected neuromuscular disease/pre-existing weakness,

Creatinine clearance less than 30 ml/min

Bradycardia of less than 40 beats/min,

Pregnancy, breast feeding women

Known or suspected allergy to BRIDION® (sugammadex), neostigmine or rocuronium.

Patients with contraindications towards sugammadex, neostigmine or rocuronium

Patients included in another trial within the last 30 days

Patients with legal guardians or surrogate decision making

Patients who refuse to use non-hormonal contraceptive method or back-up method of contraception (such as condoms and spermicides) for the next 7 days if receiving sugammadex.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 79 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavithra Ranganathan, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Healthcare Ruby Memorial Hospital, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Neostigmine: Reversal of Paralysis in Microlaryngoscopy procedures: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6-1.2 mg/kg (vitals maintained within 20% of baseline). Standard anti-nausea prophylaxis - Ondansetran and Decadran intraoperative.After induction; amount of inhaled anesthetic and remifentanil used will be titrated based on hemodynamic parameters (maintained within 20% from baseline) and a BIS monitor.TOF testing done every 5 minutes:Group 1 will receive reversal with neostigmine (0.04 mg/kg and glycopyrrolate (0.01 mg/kg)
  neostigmine: receive reversal with neostigmine 0.04 mg/kg
  glycopyrrolate: receive reversal with glycopyrrolate (0.01 mg/kg)
- Group 2 Sugammadex: Reversal of Paralysis in Microlaryngoscopy procedures: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6-1.2 mg/kg (vitals maintained within 20% of baseline). Standard anti-nausea prophylaxis - Ondansetran and Decadran intraoperative.After induction; amount of inhaled anesthetic and remifentanil used will be titrated based on hemodynamic parameters (maintained within 20% from baseline) and a BIS monitor.TOF testing done every 5 minutes: Group2 will receive reversal with sugammadex 4mg/kg
  Sugammadex: receive reversal with sugammadex 4mg/kg
Period: Overall Study
Arm/Group | Group 1 Neostigmine | Group 2 Sugammadex
Started | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Neostigmine: Reversal of Paralysis in Microlaryngoscopy procedures: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6-1.2 mg/kg (vitals maintained within 20% of baseline). Standard anti-nausea prophylaxis - Ondansetran and Decadran intraoperative.After induction; amount of inhaled anesthetic and remifentanil used will be titrated based on hemodynamic parameters (maintained within 20% from baseline) and a BIS monitor.TOF testing done every 5 minutes:Group 1 will receive reversal with neostigmine (0.04 mg/kg and glycopyrrolate (0.01 mg/kg)
  neostigmine: receive reversal with neostigmine 0.04 mg/kg
  glycopyrrolate: receive reversal with glycopyrrolate (0.01 mg/kg)
- Sugammadex: Reversal of Paralysis in Microlaryngoscopy procedures: Inhaled anesthetics: sevoflurane at 1 MAC, remifentanil and intubation with rocuronium at 0.6-1.2 mg/kg (vitals maintained within 20% of baseline). Standard anti-nausea prophylaxis - Ondansetran and Decadran intraoperative.After induction; amount of inhaled anesthetic and remifentanil used will be titrated based on hemodynamic parameters (maintained within 20% from baseline) and a BIS monitor.TOF testing done every 5 minutes: Group2 will receive reversal with sugammadex 4mg/kg
  Sugammadex: receive reversal with sugammadex 4mg/kg
- Total: Total of all reporting groups
Arm/Group | Neostigmine | Sugammadex | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.62 (10.99) | 60.04 (11.41) | 59.83 (.296)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 26 | 23 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Extubation After End of Procedure
Description: West Virginia University Hospitals use an electronic medical record (EMR) to chart the end of the procedure. When the surgeon states "We are done", always at withdrawal of the scope, extubation begins. From the time we chart end of procedure to the time of extubation is the extubation time. The start and end times for extubation will be recorded in the EMR.
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 40 | 39
Minutes | 11.06 (6.51) | 10.36 (5.37)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Neostigmine | Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03111121/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03111121/ICF_001.pdf